CLINICAL TRIAL: NCT06772480
Title: Thalidomide Versus Argon Plasma Coagulation in Gastric Antral Vascular Ectasia(GAVE)-Related Anaemia in Cirrhosis (TAG Trial)- A Randomised Controlled Trial
Brief Title: Thalidomide Versus Argon Plasma Coagulation in Gastric Antral Vascular Ectasia(GAVE)-Related Anaemia in Cirrhosis (TAG Trial)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-70
Record Dates: First submitted 2025-01-01; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-12

CONDITIONS: Liver Cirrhosis; Gastric Antral Vascular Ectasia
MeSH Terms: conditions — Liver Cirrhosis; Gastric Antral Vascular Ectasia | interventions — Thalidomide; Argon Plasma Coagulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thalidomide Group (Experimental): Patients will receive oral thalidomide starting at 50 mg daily, with a weekly increase of 50 mg up to a maximum of 200 mg daily, continued for four months.
  Interventions: Drug: Thalidomide
- APC Group (Active Comparator): Patients will undergo APC treatment every 2-3 weeks initially, followed by maintenance sessions every three months as required.
  Interventions: Procedure: Argon Plasma Coagulation

INTERVENTIONS:
Drug: Thalidomide — Patients will receive oral thalidomide starting at 50 mg daily, with a weekly increase of 50 mg up to a maximum of 200 mg daily, continued for four months
  Arms: Thalidomide Group
Procedure: Argon Plasma Coagulation — Patients will undergo APC treatment every 2-3 weeks initially, followed by maintenance sessions every three months as required.
  Arms: APC Group

SUMMARY:
Gastric Antral Vascular Ectasia (GAVE) is an erosive form of gastritis distinguished by veno-capillary ectasia, which manifests as tortuous columns of dilated vessels. Histologically, these vessels show dilated mucosal capillaries filled with fibrin thrombi, accompanied by fibromuscular hyperplasia and spindle cell proliferation of the lamina propria. GAVE is prevalent in about 12% of patients with cirrhosis, with 60-70% of these patients becoming transfusion-dependent due to severe anaemia caused by GAVE related bleeding. The most commonly used treatment for GAVE is endoscopic therapy using Argon Plasma Coagulation (APC), which, while effective, often requires multiple sessions due to a high recurrence rate of 30-60%. These frequent interventions increase the burden on patients and healthcare systems. As a result, alternative treatments have been sought. Thalidomide, known for its potent antiangiogenic properties, significantly lowers vascular endothelial growth factor (VEGF) levels, offering a promising non-invasive treatment option. Early studies, such as those by García-Pagán have demonstrated thalidomide's effectiveness in reducing transfusion requirements and managing bleeding in cirrhotic patients with GAVE, yet its comprehensive efficacy and safety profile remains under-studied. This project aims to rigorously evaluate the efficacy and safety of thalidomide compared to APC in managing GAVE-related anemia in cirrhotic patients. Through a controlled trial, this study will provide vital data to potentially shift treatment paradigms, enhance patient quality of life, and reduce the need for repetitive invasive procedures.

DETAILED DESCRIPTION:
Aim: To evaluate and compare the efficacy and safety of thalidomide with argon plasma coagulation (APC) in managing gastric antral vascular ectasia (GAVE)-related anaemia in patients with cirrhosis.

Hypothesis: Thalidomide, due to its antiangiogenic effects, will more effectively reduce GAVE-related bleeding, improve haemoglobin levels, and decrease transfusion dependency compared to APC in patients with cirrhosis and GAVE-related anaemia.

Study Design:

Single-centre, open-label, randomised controlled trial to compare the efficacy and safety of thalidomide versus argon plasma coagulation (APC) in managing GAVE-related anaemia in cirrhotic patients.

Study Population:

Adult patients (aged 18-65 years) diagnosed with cirrhosis and endoscopically confirmed GAVE-related anaemia, presenting at the Institute of Liver and Biliary Sciences.

Randomization: Patients will be randomly assigned to receive either thalidomide or APC in a 1:1 ratio by block randomization method with block size of 10 and it will be implemented by using ILBS IWRS facility.

Follow-up and Assessments:

* Patients will be followed every two weeks for the first month, then monthly up to six months. Assessments will include haemoglobin levels, the number of transfused blood units, the frequency of bleeding episodes, hospitalizations, and the number of required endoscopic sessions.
* Adverse effects will be monitored and recorded at each visit.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (aged ≥18 - 65years)
2. Cirrhosis
3. Endoscopically confirmed diagnosis of GAVE

   1. +/- GAVE with active ooze
   2. Iron deficiency anemia*
4. Ability to provide informed consent

Exclusion Criteria:

1. CTP >/=13
2. Active GI Bleeding is caused by a cause other than GAVE.
3. Renal insufficiency ( Creatinine >3mg/dL and/or on RRT)
4. Pregnancy or childbearing age
5. Contraindications to thalidomide therapy: Severe peripheral neuropathy or seizures or a history of thromboembolic disease.
6. Use of antiangiogenic drugs
7. Bevacizumab, steroids, octreotide
8. Severe cardiopulmonary disorders
9. H/o thalidomide use in the past 3months
10. Contraindications to APC: Coagulopathy( Pacemaker or implantable defibrillator, Platelet <45000, INR: >1.8 )
11. Overt Hepatic Encephalopathy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-05 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Mean increase in hemoglobin levels from baseline | 4 months

SECONDARY OUTCOMES:
Atleast 50 percent change in requirement of PRBCs transfusions at the end of 4 months | 4 months
Increase in serum iron levels, percent transferrin saturation at the end of 4months | 4 months
Change in amount of PRBC's transfused at the end of 4 months. | 4 months
Change in GAVE related bleeding episodes at the end of 4 months | 4 months
Number of hospitalizations due to GAVE related anemia, in 4 months | 4 months
Duration of days of hospitalization due to GAVE related anemia in 4 months | 4 months
Need of rescue endoscopic sessions in 4 months in thalidomide group | 4 months
Endoscopic resolution of GAVE at the end of 4 months | 4 months
  Endoscopic resolution is defined as endoscopic findings of GAVE as absent.
Change in VEGF levels in Thalidomide group at the end of 4 months | 4 months
Change in pepsinogen levels in Thalidomide group at the end of 4 months | 4 months
Change in gastrin levels in Thalidomide group at the end of 4 months | 4 months
Adverse events in each group at the end of 4 months | 4 months
Quality of life measures - Short Form 36 | 4 months
  Quality of life measures - Short Form 36 ranges from 0 to 100, 0 indicate maximum disability and 100 indicate no disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences (ILBS), New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided